CLINICAL TRIAL: NCT06620107
Title: Noninvasive High Frequency Oscillation Ventilation (NHFOV) in Comparison to Noninvasive Intermittent Positive Pressure Ventilation (NIPPV) As Post-extubation Support in Preterm Neonates
Brief Title: NHFOV Vs NIPPV Post-extubation in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Wafaa Mahmoud Hassan Abouseada, pediatric demonstrator at faculty of medicine- kafrelsheikh university, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NHFOV vs NIPPV in neonates
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Noninvasive high frequency oscillation ventilation (Active Comparator): preterm neonates with GA of 32 to 36 weeks ready for extubation
  Interventions: Device: noninvasive high frequency oscillation ventilation
- Noninvasive intermittent positive pressure ventilation (Active Comparator): preterm neonates with GA of 32 to 36 weeks ready for extubation
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive high frequency oscillation ventilation — cases of group A extubated on NHFOV, and it will be provided by CNO, Medin device, Germany) via binasal prongs with the following parameters:
  * MAP of 6 cmH2O and will be titrated targeting a FiO2 ≤ 25-30%, maximum FiO2 will be 40% and target oxygen saturation will be 90-95%.
  * Frequency of 8 Hz and can be changed within the range of 8-12 Hz.
  * Amplitude of 7 cmH2O and can be titrated within the range of 7-10 cmH2O according to PaCO2.
  Arms: Noninvasive high frequency oscillation ventilation
Device: noninvasive positive pressure ventilation — NIPPV will be provided by any type of neonatal ventilator available in the unit via binasal prongs starting with the following parameters:
  * Positive end expiratory pressure (PEEP) of 5 cmH2O and can be titrated to 8 cmH2O according to the oxygenation .
  * Peak inspiratory pressure (PIP) of 15 cmH2O and can be titrated to 25 cmH2O ,according to oxygenation , PaCO2 level and the chest expansion .
  * FiO2 ≤ 25-30% and can be increased to 40 % maximally targeting oxygen saturation of 90-95% .
  * Inspiratory time of 0.40-0.50 s .
  * Rate of 30 bpm and can be increased to maximum 50 bpm .
  * Synchronization will not be applied.
  Arms: Noninvasive intermittent positive pressure ventilation

SUMMARY:
comparison between Noninvasive Intermittent Positive Pressure Ventilation (NIPPV) and Noninvasive High Frequency Oscillation Ventilation (NHFOV) post-extubation in preterm neonates as regards the efficacy and their possible complications.

DETAILED DESCRIPTION:
The global definition of preterm infant by the World Health Organization is any infant born before 37 weeks of gestation. Annually, an estimated 15 million (11.1%) preterm infants are born worldwide. Preterm birth is further classified as extremely preterm (<28 weeks), very preterm (28 to <32 weeks), and moderate (32 to <34 weeks) to late preterm (34 to <37 weeks).

Prematurity has been associated with several risk factors, such as history of previous preterm birth, pregnancy induced hypertension, premature rupture of fetal membranes, multiple pregnancy, bleeding during pregnancy, history of abortion, fetal malformation, inadequate antenatal care, polyhydramnios and previous caesarean section.

Preterm neonates are at greater risk of a range of short-term and long-term morbidities. Respiratory distress syndrome (RDS) is one of the most common causes of morbidity and mortality in preterm infants. RDS is characterized by a lack of lung surfactant. Insufficient surfactant production or secretion results in higher alveolar surface tension, leading to atelectasis and impaired gas exchange. Respiratory distress typically manifests in newborns as tachypnea, intercostal retractions, nasal flaring, grunting, and cyanosis.

Invasive mechanical ventilation (IMV) increases survival in preterm infants with severe RDS. However, prolonged intubation and mechanical ventilation of preterm infants increases the risk of life-threatening complications including, ventilator induced lung injury and airway inflammation leading to bronchopulmonary dysplasia, and nosocomial pneumonia, and also increases the risk of a poor neurodevelopmental outcome. Therefore, when caring for premature infants, clinicians should focus on weaning from IMV as expeditiously as possible to noninvasive respiratory support (NRS).

There are many strategies and criteria for weaning, including evaluation of ventilatory parameters, clinical/biochemical criteria, and predictive indices of extubation that can be followed by or combined with spontaneous breathing trials or gradual withdrawal from ventilatory support.

Noninvasive respiratory support modalities include continuous positive airway pressure (CPAP), high flow nasal cannula (HFNC), noninvasive intermittent positive pressure ventilation (NIPPV), bilevel CPAP (BiPAP) and noninvasive high frequency oscillation ventilation (NHFOV).

NIPPV is a time cycled, pressure limited mode of ventilation. Conventional ventilator is used to generate two levels of pressures, namely, Peak inspiratory pressure and positive end expiratory pressure. Additionally, a backup rate is provided typically using longer inspiratory time. The main drawback of neonatal NIPPV is the lack of synchronization, which is difficult to achieve and is often unavailable.

NHFOV is the application of a bias flow generating a continuous distending positive pressure with superimposed oscillations which have a constant frequency and an active expiratory phase. NHFOV combines the advantages of NCPAP and high-frequency ventilation, making it more effective at maintaining alveolar stability, eliminating CO2, and limiting barotrauma.

The study assumed that NHFOV is more efficacious than NIPPV as regard prevention of the need for re-intubation in preterm infants with gestational age between 32 and 36 weeks and 6 days after their 1st extubation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age between 32 and 36 weeks and on mechanical ventilation ready to be extubated.

When the case is ready for extubation , will receive at least one loading dose of caffeine citrate (20 mg/kg/dose) and daily maintenance dose of 5 mg/kg/dose.

Criteria for extubation:

* Blood gas analysis: PH > 7.25 and PaCO2 ≤ 60 mmHg.
* Airway pressure (Paw) of 7 to 8 cmH2O.
* Required fraction of inspired oxygen (FiO2) ≤ 30%.
* Sufficient spontaneous breathing by clinical evaluation.

Exclusion Criteria:

* Full term neonates.
* Preterm neonates who will not require intubation.
* Preterm neonates with one of the following criteria:

birth weight > 900 gms , major congenital anomalies, upper airway anomalies, neuromuscular diseases, surgical cases, intraventricular hemorrhage grade IV.

• Cases that require reintubation after more than 72 hours of extubation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
reintubation and the duration of respiratory support | from the date of birth till the date of discharge from NICU or death (assessed up to 3 months)..
  * The number of cases that required re-intubation and the time of failure of extubation in hours.
  * Duration of different types of respiratory support since birth till discharge from NICU.

SECONDARY OUTCOMES:
complications | from the date of birth till the date of discharge from NICU or death (assessed up to 3 months).
  * Airleak syndromes.
  * Apnea rate.
  * Nasal septal injury.
  * Bronchopulmonary dysplasia.
  * Intraventricular hemorrhage ≥ 2nd grade.
  * Hemodynamically significant PDA.
  * Retinopathy of prematurity ≥ 2nd stage.
  * Necrotizing enterocolitis ≥ 2nd stage.
  * Frequency of vomiting.
  * Feeding intolerance.
  * Weekly weight gain until NICU discharge.
  * Duration of hospitalization.
  * Mortality during stay in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Heba SM El-Mahdy, Study Chair — Tanta University
Locations (1):
- Kafrelsheikh University, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi Y, Muniraman H, Biniwale M, Ramanathan R. A Review on Non-invasive Respiratory Support for Management of Respiratory Distress in Extremely Preterm Infants. Front Pediatr. 2020 May 28;8:270. doi: 10.3389/fped.2020.00270. eCollection 2020. PMID 32548084
- See also: Noninvasive high-frequency oscillatory ventilation versus nasal continuous positive airway pressure in preterm infants with moderate-severe respiratory distress syndrome: A preliminary report — https://pubmed.ncbi.nlm.nih.gov/28672094